CLINICAL TRIAL: NCT04950881
Title: Ultrasound-guided Cervical Vagus Nerve Block Prevents Ocularvagal Reflex in Ophthalmic Surgery
Brief Title: Cervical Vagus Nerve Block Prevents Ocularvagal Reflex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Qingxiang Mao, professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-55
Record Dates: First submitted 2021-06-20; First posted 2021-07-06 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Reflex, Oculocardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Conventional monitor and treatment The surgery is performed after patient is under general anesthesia. If patient's heart rate significantly slows down or bradycardia/arrhythmia happens, the surgeon will be asked to suspend the operation. Meanwhile, atropine (0.01-0.02mg/kg) is given intravenously to increase the heart rate. If atropine fails to increase the heart rate, isoproterenol (1-2 μg/per time) will be given intravenously to increase the heart rate.
  Interventions: Drug: Bradycardia Treatment
- Nerve block group (Experimental): After the patient is under general anesthesia, an attending physicians perform the ultrasound-guided cervical vagus nerve block (using a 50mm Braun nerve stimulation needle, and the patients were injected with 10ml of lidocaine or ropivacaine ). Then the operation starts. If patient's heart rate significantly slows down or bradycardia/arrhythmia happens, the surgeon will be asked to suspend the operation. Meanwhile, atropine (0.01-0.02mg/kg) is given intravenously to increase the heart rate. If atropine fails to increase the heart rate, isoproterenol (1-2 μg/per time) will be given intravenously to increase the heart rate. After endotracheal tube is removed, the patient will be followed up for next 24 hours.
  Interventions: Procedure: Ultrasound guided vagus nerve block; Drug: Bradycardia Treatment

INTERVENTIONS:
Procedure: Ultrasound guided vagus nerve block — Before the operation starts, patients received the ultrasound guided vagus nerve block. A 50mm Braun nerve stimulation needle is guided by the ultrasonic beam to insert into the carotid sheath and 10ml of lidocaine or ropivacaine is injected.
  Arms: Nerve block group
Drug: Bradycardia Treatment — If the OVR happens because the surgical stimulation, the operation suspends and atropine (0.01-0.02mg/kg) or isoproterenol (1-2 μg/per time)is given intravenously to increase the heart rate.

SUMMARY:
In ophthalmic surgery, surgical operations such as pulling certain eye tissues or compressing the eyeball often leads to bradycardia, arrhythmia even cardiac arrest, bradypnea, nausea and vomiting and elevated blood sugar level. The condition is called the ocularvagal reflex (OVR). Traditionally, when the bradycardia or arrhythmia happens, the operation has to be suspended, and atropine or isoproterenol is given intravenously to treat the bradycardia. Vagus nerve block may be an effective way to prevent and alleviate this vagal reflex. However it is difficult to perform the nerve block with anatomical landmark (blind) methods. In this study, the investigators used ultrasound-guided right cervical vagus nerve block to reduce the incidence of the OVR. The researchers hypothesized that low concentrations of lidocaine or ropivacaine can block the right cervical vagus nerve and reduce the incidence of intraoperative OVR. Researchers evaluated the changes of heart rate, blood pressure, oxygen saturation, and airway pressure in patients undergoing high-risk OVR surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients received surgeries with high-risk OVR, including the strabismus surgery, the posterior scleral reinforcement, and the insertion of ocular implant.

Exclusion Criteria:

* Those who have pre-existed vocal cord damage before surgery (such as hoarseness, electronic laryngoscopy shows fixed vocal cords or arytenoid cartilage dislocation).
* Those with a history of surgery on the both sides of the neck (eg, thyroidectomy, carotid endarterectomy).
* American Society of Anesthesiologist (ASA) Grade > 3
* Patients with infection at the neck puncture site, or severe coagulation abnormalities before surgery, or a history of local anesthetic allergy, or who have a pacemaker.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes of heart rate | during the operation
  Changes of heart rate in beat per minute from Baseline

SECONDARY OUTCOMES:
Changes of Blood pressure | during the operation
  Changes of systolic blood pressure in mmHg from Baseline
Changes of Peak airway pressure | during the operation
  Changes of Blood pressure in mmHg from Baseline
Changes of SpO2 | during the operation
  Changes of SpO2 in percentage in mmHg from Baseline
Nausea and vomiting in times | 24 hours after the operation
Voice changes in grades (0-3) | 24 hours after the operation
  Changes of Voice changes in grades (0-3) from Baseline. 0 means good, 2 means moderate change of voice, 3 means hoarse voice

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Army Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Casutt M, Breitenmoser I, Werner L, Seelos R, Konrad C. Ultrasound-guided carotid sheath block for carotid endarterectomy: a case series of the spread of injectate. Heart Lung Vessel. 2015;7(2):168-176. PMID 26157743
- [Background] Arnold RW, Bond AN, McCall M, Lunoe L. The oculocardiac reflex and depth of anesthesia measured by brain wave. BMC Anesthesiol. 2019 Mar 14;19(1):36. doi: 10.1186/s12871-019-0712-z. PMID 30871507